CLINICAL TRIAL: NCT03024671
Title: Epicutaneous Testing of Cosmetic Products to Determine Skin Compatibility
Brief Title: Epicutaneous Testing of Cosmetics for Skin Compatibility
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Mibelle AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KEK-BE 2016-01686
Record Dates: First submitted 2017-01-11; First posted 2017-01-19 (Estimated); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Dermatitis
MeSH Terms: conditions — Dermatitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patch test (Experimental): Patients with patch test of cosmetics
  Interventions: Other: Patch test application

INTERVENTIONS:
Other: Patch test application — test patch with cosmetic product will be applied to the back

SUMMARY:
The dermatological testing of cosmetic products which are new on the market, or existing products with novel formulations is common and a useful procedure, yet necessary to alleviate common irritants and contact allergic reactions. Cosmetic products contain a range of substances that may be considered as potential irritants or contact allergens. In order to estimate that risk, cosmetics are tested by applying patch tests.

DETAILED DESCRIPTION:
The dermatological testing of cosmetic products which are new on the market, or existing products with novel formulations is common and a useful procedure, yet necessary to alleviate common irritants and contact allergic reactions. Cosmetic products contain a range of substances that may be considered as potential irritants or contact allergens. In order to estimate that risk, cosmetics are tested by applying patch tests, as with allergic reactions.

ELIGIBILITY:
Inclusion Criteria:

* Men and women older than 18 years old
* Persons undergoing a diagnostic patch test for reason of a skin disease
* Signed written informed consent

Exclusion Criteria:

* Acute skin inflammation and eczema on the back
* Systemic corticosteroid and immunosuppressive therapy as well as UV exposure of the back within the last 4 weeks
* Topical corticosteroids used on the back within the last two weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-02-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with positive patch test reactions to cosmetics | 4 weeks
  Inflammation of Skin at test patch location

CONTACTS AND LOCATIONS:
Overall Officials: Dagmar Simon, MD, Principal Investigator — Dept. of Dermatology, Inselspital
Locations (1):
- Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
single centered study